CLINICAL TRIAL: NCT04782518
Title: Personalizing Exercise for Parkinson Disease
Acronym: PEP
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202002075
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: exercise; physical activity
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with PD: Adults with Parkinson Disease. This is an observational study without an intervention.

SUMMARY:
The overarching aim is to determine the benefits of Parkinson-specific exercise programs and general exercise patterns on physical function and disease-related quality of life among people with Parkinson Disease (PD). The significance of this project is that millions of individuals experience adverse consequences of PD and there is strong evidence that structured exercise programs have beneficial effects on motor function and PD-related quality of life. Participation in this study involves online surveys upon enrollment (i.e., baseline) and at 3 months, 6 months, 9 months, 1 year, and 2 years.

DETAILED DESCRIPTION:
Parkinson Disease (PD) is a neurodegenerative disease that affects more than ten million people worldwide. In the United States, more than one million people are living with PD and more than 100,000 new cases are diagnosed each year.

Exercise to Ease the Burden of PD:

Exercise is an adjunct to pharmacologic therapy for PD that has been shown in many intensive research studies to help improve motor and non-motor symptoms in PD. A variety of Parkinson-specific exercise programs have been developed to help improve balance, posture, mobility, strength, endurance, speech, and/or self-help skills. These classes include various modes of exercise and different intensity levels, tailored for patients' personal characteristics and functional abilities.

Current Gaps in Knowledge and Aim:

The benefits of PD-specific exercise programs on physical function and disease-related quality of life have not been evaluated. Furthermore, many patients may not have access to PD-specific exercise programs. The proposed project addresses these gaps by exploring associations between PD-specific exercise programs and several metrics of physical function and quality of life among individuals with PD. In addition, the investigators are studying associations among overall exercise patterns, physical activity patterns, physical function, and quality of life among individuals with PD.

Study Involvement:

Participation in this study involves online surveys completed upon enrollment (i.e., baseline) and at 3 months, 6 months, 9 months, 1 year, and 2 years. A family member, caregiver, or friend may help the participant complete the online surveys.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson Disease
* Ability to provide informed consent

Exclusion Criteria:

* Children (<18 years of age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have been diagnosed by a physician as having Parkinson Disease are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Association between exercise patterns and quality of life | Baseline
  Association between exercise patterns (including exercise type and frequency) and quality of life, as assessed by the Parkinson's Disease Questionnaire (PDQ-39). The score range for the PDQ-39 is 0 to 100, with lower scores reflecting higher quality of life.
Association between exercise patterns and mobility | Baseline
  Association between exercise patterns (including exercise type and frequency) and mobility, as assessed by the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire. The Neuro-QOL short form domain on Lower Extremity Function - Mobility will be used. The score range for the Neuro-QOL Mobility domain is 8 to 40, with higher scores reflecting a higher level of lower extremity function and mobility (i.e., better self-reported health).
Association between exercise patterns and well-being | Baseline
  Association between exercise patterns (including exercise type and frequency) and well-being, as assessed by the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire. The Neuro-QOL short form domain on Positive Affect and Well-Being will be used. The score range for the Neuro-QOL Positive Affect and Well-Being domain is 9 to 45, with higher scores reflecting a higher level of well-being.
Association between exercise patterns and quality of life | 2 years
  Association between exercise patterns (including exercise type and frequency) and quality of life, as assessed by the Parkinson's Disease Questionnaire (PDQ-39). The score range for the PDQ-39 is 0 to 100, with lower scores reflecting higher quality of life.
Association between exercise patterns and mobility | 2 years
  Association between exercise patterns (including exercise type and frequency) and mobility, as assessed by the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire. The Neuro-QOL short form domain on Lower Extremity Function - Mobility will be used. The score range for the Neuro-QOL Mobility domain is 8 to 40, with higher scores reflecting a higher level of lower extremity function and mobility (i.e., better self-reported health).
Association between exercise patterns and well-being | 2 years
  Association between exercise patterns (including exercise type and frequency) and well-being, as assessed by the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire. The Neuro-QOL short form domain on Positive Affect and Well-Being will be used. The score range for the Neuro-QOL Positive Affect and Well-Being domain is 9 to 45, with higher scores reflecting a higher level of well-being.

SECONDARY OUTCOMES:
Proportion of participants who attend a PD-specific exercise class | Baseline
  Number of participants who attend a PD-specific exercise class relative to the total number of study participants.
Frequency of participation in exercise classes or recreational exercise | Baseline
  Frequency distribution of participation in exercise classes or recreational exercise, expressed on a weekly basis.
Quality of Life score on the Parkinson's Disease Questionnaire (PDQ-39) | Baseline
  Quality of Life summary index score on the Parkinson's Disease Questionnaire (PDQ-39). The score range for the PDQ-39 is 0 to 100, with lower scores reflecting higher quality of life.
Mobility score on the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire | Baseline
  Mobility score will be computed from the Quality of Life in Neurological Disorders (Neuro-QOL) short form questionnaire. The Neuro-QOL short form domain on Lower Extremity Function - Mobility will be used. The score range for the Neuro-QOL Mobility domain is 8-40, with higher scores reflecting a higher level of lower extremity function and mobility (i.e., better self-reported health).
Well-being score on the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire | Baseline
  Well-being will be assessed by the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire. The Neuro-QOL short form domain on Positive Affect and Well-Being will be used. The score range for the Neuro-QOL Positive Affect and Well-Being domain is 9 to 45, with higher scores reflecting a higher level of well-being.
Proportion of participants who attend a PD-specific exercise class | 2 years
  Number of participants who attend a PD-specific exercise class relative to the total number of study participants.
Frequency of participation in exercise classes or recreational exercise | 2 years
  Frequency distribution of participation in exercise classes or recreational exercise, expressed on a weekly basis.
Quality of Life score on the Parkinson's Disease Questionnaire (PDQ-39) | 2 years
  Quality of Life summary index score on the Parkinson's Disease Questionnaire (PDQ-39). The score range for the PDQ-39 is 0 to 100, with lower scores reflecting higher quality of life.
Mobility score on the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire | 2 years
  Mobility score will be computed from the Quality of Life in Neurological Disorders (Neuro-QOL) short form questionnaire. The Neuro-QOL short form domain on Lower Extremity Function - Mobility will be used. The score range for the Neuro-QOL Mobility domain is 8-40, with higher scores reflecting a higher level of lower extremity function and mobility (i.e., better self-reported health).
Well-being score on the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire | 2 years
  Well-being will be assessed by the Quality of Life in Neurological Disorders (Neuro-QOL) questionnaire. The Neuro-QOL short form domain on Positive Affect and Well-Being will be used. The score range for the Neuro-QOL Positive Affect and Well-Being domain is 9 to 45, with higher scores reflecting a higher level of well-being.

OTHER OUTCOMES:
Age of participants (in years) | Baseline
  Age of participants (years)
Proportion of men and women | Baseline
  Number of men and number of women relative to the total number of study participants
State or country of residence | Baseline
  State of residence (for those living in the United States) or country of residence (for those living outside the United States)
Year of diagnosis of Parkinson Disease | Baseline
  Year in which the participant was diagnosed as having Parkinson Disease
Proportion of participants who tested positive for coronavirus | Baseline
  Number of participants who tested positive for coronavirus relative to the total number of study participants. Coronavirus is the virus that causes coronavirus disease 2019 (COVID-19).
Proportion of participants who have received a vaccine for coronavirus disease 2019 (COVID-19) | Baseline
  Number of participants who have received a vaccine for coronavirus disease 2019 (COVID-19) relative to the total number of study participants.
Proportion of participants who do not intend to receive a vaccine for coronavirus disease 2019 (COVID-19) | Baseline
  Number of participants who do not intend to receive a vaccine for coronavirus disease 2019 (COVID-19) relative to the total number of study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Racette, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Aggregate data that contains no HIPPA identifiers will be made available as required if the request complies with all federal and Washington University School of Medicine policies for data sharing. Individual participant data (IPD) that may be shared include standardized survey scores, such as the Parkinson's Disease Questionnaire - 39 (PDQ-39) single index score, the PDQ-39 subscores, the Quality of Life in Neurological Disorders (Neuro-QoL) Lower Extremity Function - Mobility score, and the Neuro-QoL Positive Affect and Well-Being score. Any individual-level data that are shared will be de-identified.

REFERENCES:
- [Background] Wright Willis A, Evanoff BA, Lian M, Criswell SR, Racette BA. Geographic and ethnic variation in Parkinson disease: a population-based study of US Medicare beneficiaries. Neuroepidemiology. 2010;34(3):143-51. doi: 10.1159/000275491. Epub 2010 Jan 15. PMID 20090375
- [Background] Nadeau A, Pourcher E, Corbeil P. Effects of 24 wk of treadmill training on gait performance in Parkinson's disease. Med Sci Sports Exerc. 2014 Apr;46(4):645-55. doi: 10.1249/MSS.0000000000000144. PMID 24002341
- [Background] Ramaswamy B, Jones J, Carroll C. Exercise for people with Parkinson's: a practical approach. Pract Neurol. 2018 Oct;18(5):399-406. doi: 10.1136/practneurol-2018-001930. Epub 2018 Jun 1. PMID 29858216
- [Background] Rossi A, Torres-Panchame R, Gallo PM, Marcus AR, States RA. What makes a group fitness program for people with Parkinson's disease endure? A mixed-methods study of multiple stakeholders. Complement Ther Med. 2018 Dec;41:320-327. doi: 10.1016/j.ctim.2018.08.012. Epub 2018 Aug 31. PMID 30477861
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479
- [Background] Fitzpatrick R, Jenkinson C, Peto V, Hyman N, Greenhall R. Desirable properties for instruments assessing quality of life: evidence from the PDQ-39. J Neurol Neurosurg Psychiatry. 1997 Jan;62(1):104. doi: 10.1136/jnnp.62.1.104. No abstract available. PMID 9010413
- [Background] Jenkinson C, Peto V, Fitzpatrick R, Greenhall R, Hyman N. Self-reported functioning and well-being in patients with Parkinson's disease: comparison of the short-form health survey (SF-36) and the Parkinson's Disease Questionnaire (PDQ-39). Age Ageing. 1995 Nov;24(6):505-9. doi: 10.1093/ageing/24.6.505. PMID 8588541
- [Background] Peto V, Jenkinson C, Fitzpatrick R, Greenhall R. The development and validation of a short measure of functioning and well being for individuals with Parkinson's disease. Qual Life Res. 1995 Jun;4(3):241-8. doi: 10.1007/BF02260863. PMID 7613534
- [Background] Peto V, Jenkinson C, Fitzpatrick R. Determining minimally important differences for the PDQ-39 Parkinson's disease questionnaire. Age Ageing. 2001 Jul;30(4):299-302. doi: 10.1093/ageing/30.4.299. PMID 11509307
- [Background] Harrison JE, Preston S, Blunt SB. Measuring symptom change in patients with Parkinson's disease. Age Ageing. 2000 Jan;29(1):41-5. doi: 10.1093/ageing/29.1.41. PMID 10690694